CLINICAL TRIAL: NCT03681132
Title: The Norwegian Nucleoside Analogue Stop Study: a Randomized Open-label Trial in HBeAg Negative Chronic Hepatitis B, Aiming at Achieving a Functional Cure.
Brief Title: The Norwegian Nucleoside Analogue Stop Study
Acronym: Nuc-Stop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Addis Ababa University (Other); St. Paul's Hospital Millennium Medical College, Ethiopia (Other); South-Eastern Norway Regional Health Authority, Norway (Unknown); Bærum Hospital, Norway (Unknown); Drammen Hospital, Norway (Unknown); Tønsberg Hospital, Norway (Unknown); Helse Stavanger HF (Other Government); Ålesund Hospital, Norway (Unknown); Bodø Hospital, Norway (Unknown); Hvidovre University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Asgeir Johannessen, Consultant/ researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/988
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-threshold re-start (Other): Re-start antiviral therapy if HBV DNA viral load >2000 IU/ml and ALT >80 U/L.
  Interventions: Other: Stop of therapy
- High-threshold re-start (Other): Re-start antiviral therapy if:
  * ALT >100 U/L persisting for more than 4 months without any spontaneous decline toward normal; OR
  * ALT >400 U/L persisting for more than 2 months in consecutive assays.
  Interventions: Other: Stop of therapy

INTERVENTIONS:
Other: Stop of therapy — The active intervention is to stop antiviral therapy, and delay re-start in the high-threshold group.

SUMMARY:
Globally, an estimated 257 million individuals have chronic hepatitis B-virus infection (CHB). In the absence of treatment 15-40% of these will progress to liver cirrhosis and/or hepatocellular carcinoma. Oral antiviral treatment suppresses the virus and improves prognosis, but less than 0.5% per year achieve a "functional cure" (i.e. HBsAg loss). One remaining controversy, therefore, is whether antiviral treatment must continue life-long. Observational studies have assessed stopping antiviral treatment after years of viral suppression; however, HBsAg loss has rarely been seen. But interestingly, a few small trials that chose watchful waiting instead of re-initiation of treatment when reactivation occurred, achieved 40% HBsAg loss during 6 years follow-up.

The present proposal is a randomized controlled trial that will assess the safety, efficacy, and cost-effectiveness of treatment discontinuation - and delayed restart - in HBeAg negative CHB. The study is sufficiently powered to address the hypotheses, and a pilot study that demonstrates feasibility has been performed. Patients will be enrolled at 12 Norwegian hospitals, in addition to our collaborating institution in Ethiopia - the largest CHB treatment center in sub-Saharan Africa. If the study shows that discontinuation is safe and effective, it will directly impact both national and international treatment guidelines.

Main objective:

-To study whether stopping nucleoside analogue (NA) therapy - and delaying re-start - can trigger an immune response and set off a functional cure (viz HBsAg loss)

Secondary objectives:

* Assess whether stopping NA therapy - and delaying re-start - leads to a higher chance of HBsAg loss
* Assess the safety of stopping NA therapy - and delaying re-start - in terms of hepatic decompensation, fibrosis progression, and/or adverse events
* Study whether stopping NA therapy - and delaying re-start - leads to a higher chance of sustained off-therapy immune control (low viral load and normal ALT)
* Assess the quality of life and cost-effectiveness of stopping NA therapy - and delaying re-start
* Identify predictors of HBsAg loss

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-70 years) with HBeAg negative chronic hepatitis B
* HBeAg negative at start of antiviral therapy
* Treated minimum 2 years with either tenofovir or entecavir without interruption (i.e. no self-reported episodes of ≥2 weeks off therapy)
* Full viral suppression >2 years: at least 3 measurements at least 6 months apart with at least 24 months between the first and last measurement.
* Most recent liver fibrosis assessment, performed within the past 12 months, does not show advanced fibrosis (i.e. Metavir score <F3 or Fibroscan <9 kPa). For the (few) patients who lack pre-treatment fibrosis assessment, a more conservative Fibroscan threshold of <8 kPa will apply.

Exclusion Criteria:

* A history of decompensated liver disease, either by clinical signs (ascites, encephalopathy, portal hypertension, jaundice) or suggestive laboratory results (total bilirubin >38 umol/L, INR >1.5, platelets <75,000/mm3, serum albumin <30 g/L).
* Any previous diagnosis of cirrhosis, either by liver biopsy (Metavir score F4) or elastography (Fibroscan >12 kPa). Elastography results with concomitant ALT >200 U/L are not considered.
* Previous hepatocellular carcinoma (HCC).
* Co-infections with HIV, hepatitis C or hepatitis D.
* Other disease or medication that can interfere with the study (e.g. ongoing alcohol or illicit drug abuse, immunosuppressive medication, other active liver disease, or any other condition which in the opinion of the physician is incompatible with participation)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
HBsAg loss | Within 3 years after stopping therapy
  Undetectable HBsAg measured by a standard assay

SECONDARY OUTCOMES:
Time to HBsAg loss | Within 3 years after stopping therapy
  Time from randomization to undetectable HBsAg
Time to re-start of antiviral therapy | Within 3 years after stopping therapy
  Time from randomization to re-start of therapy according to the specified criteria
Severe unintended medical events | Within 3 years after stopping therapy
  Liver failure or other liver-related grade 4/5 SAEs
Immune control | Within 3 years after stopping therapy
  Sustained off-therapy response viz HBV DNA <2000 IU/ml and ALT <40 U/L
Changes in health-related quality of life | Within 3 years after stopping therapy
  Changes in the EuroQol standardized measure of health status (EQ-5D-5L) score. The summary index (from 0 to 1) as described by the manufacturer (euroqol.org) will be employed.
Liver fibrosis evolution | Within 3 years after stopping therapy
  Changes in transient elastography from baseline

CONTACTS AND LOCATIONS:
Locations (11):
- Hvidovre Hospital, Copenhagen, Denmark
- St Paul Hospital Millennium Medical College, Addis Ababa, Ethiopia
- Norway (8):
  - Ålesund Hospital, Ålesund
  - Bodø Hospital, Bodø
  - Drammen Hospital, Drammen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Bærum Hospital, Sandvika
  - Stavanger University Hospital, Stavanger
  - Tønsberg Hospital, Tønsberg
- Karonlinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Johannessen A, Reikvam DH, Aleman S, Berhe N, Weis N, Desalegn H, Stenstad T, Heggelund L, Samuelsen E, Karlsen LN, Lindahl K, Pettersen FO, Iversen J, Kleppa E, Bollerup S, Winckelmann AA, Brugger-Synnes P, Simonsen HE, Svendsen J, Kran AB, Holmberg M, Olsen IC, Rueegg CS, Dalgard O. Clinical trial: An open-label, randomised trial of different re-start strategies after treatment withdrawal in HBeAg negative chronic hepatitis B. Aliment Pharmacol Ther. 2024 Aug;60(4):434-445. doi: 10.1111/apt.18147. Epub 2024 Jul 5. PMID 38970293
- [Derived] Holmberg M, Aass HCD, Dalgard O, Samuelsen E, Sun D, Bjorkstrom NK, Johannessen A, Reikvam DH. Treatment cessation in HBeAg-negative chronic hepatitis B: clinical response is associated with increase in specific proinflammatory cytokines. Sci Rep. 2023 Dec 18;13(1):22590. doi: 10.1038/s41598-023-50216-y. PMID 38114718